CLINICAL TRIAL: NCT06556615
Title: Development and Validation of a Standardized Assessment Instrument for Health-related Quality of Life (HrQoL) in Patients With Classical Homocystinuria
Brief Title: Health Related Quality of Life (HrQoL) in Classical Homocystinuria (CBS Deficiency)
Acronym: CBS_HrQoL
Status: Recruiting | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: CBS_HrQol
Record Dates: First submitted 2024-08-05; First posted 2024-08-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Homocystinuria
MeSH Terms: conditions — Homocystinuria | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Interview — Interviews, presentation of questionnaires

SUMMARY:
Patients, parents of young / handicapped patients, and experts will be interviewed to collect contents relevant for HrQoL in CBS deficiency. Based on these data, a questionnaire will be developed and tested for comprehensibility in patients and parents of young / handicapped patients. A final questionnaire version will be tested for psychometric criteria including validity and reliability.

ELIGIBILITY:
Inclusion criteria

* Patients with CBS deficiency from age 8 years
* Parents of patient(s) < 18 years with cognitive impairment
* Parents of patients between age 4 and 7
* Experts on CBS deficiency
* Able to give informed consent as documented by signature

Exclusion criteria

- Sufficient command of the German or the English language

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CBS deficiency from age 8 years
  * Parents of patient(s) < 18 years with cognitive impairment
  * Parents of patients between age 4 and 7
  * Experts on CBS deficiency
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
HrQol | through study completion, an average of 6 months
  Hrqol

CONTACTS AND LOCATIONS:
Locations (1):
- Kinderspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No